CLINICAL TRIAL: NCT00153712
Title: A Prospective Cohort Study to Study the Natural History and Ulcer Recurrence Without Acid Suppression of Non-NSAID, Non-HP Bleeding Peptic Ulcer Patients
Brief Title: Natural History of Non-steroidal Anti-inflammatory Drug and Non-Helicobacter Pylori in Bleeding Peptic Ulcers
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Other Study IDs: NNH Study
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Peptic Ulcer
Keywords: Non-NSAID; Non-Hp Bleeding Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non NSAID non-Hp: Patient of history of peptic ulcer bleeding with Hp-ve and without prior history of taking NSAID or Aspirin within 30 days
- Helicobacter pylori +ve: Patient with Hp+ve at peptic ulcer bleeding

SUMMARY:
The aim of this study is to study the natural history of the ulcer healing while on proton pump inhibitors (PPI) and the ulcer recurrence without acid suppression therapy of Non-steroidal Anti-inflammatory Drugs (NSAID), non-Helicobacter pylori (HP) bleeding ulcer patients.

DETAILED DESCRIPTION:
Non-steroidal Anti-inflammatory Drugs (NSAID), Non-Helicobacter pylori (HP) bleeding peptic ulcers are relatively common in the West (11%-44%). It is uncommon in Hong Kong (4%). Significant number of these patients with non-NSAID, non-Hp bleeding ulcers had co-morbid illness and many had life-threatening conditions. Our recent study showed that there is an increasing incidence of non-steroidal anti-inflammatory drugs (NSAID), non-Helicobacter pylori (Hp) bleeding peptic ulcers. There is no datum on the natural course of these patients and this is our aim to have this observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has non-NSAID (non-steroidal anti-inflammatory drugs), non-Helicobacter pylori bleeding peptic ulcer
* Age > 18 years old
* Informed consent

Exclusion Criteria:

* Concommitant use of high dose steroid or warfarin
* New start on non-steroidal anti-inflammatory drugs or aspirin or COX2 inhibitors
* Renal failure (serum creatinine > 200umol/l)
* Previous gastric surgery
* Oesophagitis, esophageal varices
* Terminal illness or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All peptic ulcer bleeding patients
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2002-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Recurrent ulcer bleeding | During the observation period
  Hematemesis or melena documented by the admitting physician, or a decrease in the hemoglobin level of at least 2 g/dL, with ulcers or bleeding erosions confirmed on endoscopy.

SECONDARY OUTCOMES:
All-cause mortality | During the observation period
  The secondary endpoint is recurrent lower gastrointestinal (GI) bleeding, which was defined as recurrent overt bleeding (melena or hematochezia without an upper GI source) or a drop in hemoglobin >2 g/dL, without an upper GI source or other non-GI causes of anemia. We excluded hemorrhoidal bleeding and colorectal cancer as lower GI outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Francis K Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Shatin, Hong Kong, China